CLINICAL TRIAL: NCT01243515
Title: Clinical Validation of a Non-Invasive Central Venous Pressure Device in Comparison With Physical Examination in Patients With Chronic Kidney Disease and Healthy Volunteers
Brief Title: Comparison of a Non-Invasive Central Venous Pressure Device and Physical Examination in Patients With Chronic Kidney Disease
Status: Withdrawn | Type: Observational
Sponsor: Mespere Lifesciences Inc. (Industry)
Collaborators: St. Joseph's Healthcare Hamilton (Other)
Responsible Party: Sponsor
Other Study IDs: MLS STP-9000006
Record Dates: First submitted 2010-11-17; First posted 2010-11-18 (Estimated); Last update posted 2013-02-08 (Estimated); Status verified 2013-02

CONDITIONS: Central Venous Pressure
Keywords: Central Venous Pressure; Kidney Diseases; Chronic Kidney Disease; Healthy Subjects; Non-Invasive Monitor
MeSH Terms: conditions — Kidney Diseases; Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Chronic Kidney Disease: minimum 7 subjects (male and female)
  Interventions: Device: Non-Invasive Central Venous Pressure monitor; Procedure: Physical examination of jugular vein
- Healthy subjects: minimum 3 subjects (male and female)
  Interventions: Device: Non-Invasive Central Venous Pressure monitor; Procedure: Physical examination of jugular vein

INTERVENTIONS:
Device: Non-Invasive Central Venous Pressure monitor — An adhesive patch (connected to the Mespere NICVP monitor) is placed on the neck of the subject, to determine if the CVP values displayed by the device correlates with CVP values obtained by physical examination (standard clinical practice)
  Other Names: NICVP monitor
Procedure: Physical examination of jugular vein — Physicians assess CVP using the jugular vein of the subject

SUMMARY:
The primary objective of this study is to determine whether a correlation exists between the Mespere Non-Invasive Central Venous Pressure (NICVP) device for measuring central venous pressure (CVP), and assessment of CVP via physical examination.

DETAILED DESCRIPTION:
The estimation of central venous pressure (CVP) is part of routine clinical examination. Central venous pressure is the indication of the pressure in the right atrium of the heart and it can be measured by determining the height of the blood column in the internal or external jugular vein. Clinical use of CVP has a wide range of applications including diagnosis of heart failure, pleural effusion, hypervolemia, hypovolemia, and sepsis. The standard clinical method for attaining CVP non-invasively is the physical examination of jugular venous pulse (JVP). The JVP provides a useful estimate of the CVP.

It is often difficult to identify the internal jugular vein to determine the JVP. The internal jugular vein is deep and adjacent to the carotid artery and pulsations derived from the artery may obscure the subtle venous pulsations. Manoeuvres to differentiate carotid pulsation and jugular pulsation are helpful in identifying the internal jugular vein, however determining the JVP based on the internal jugular vein examination is difficult.

Examination of the external jugular vein to determine JVP is an appealing alternative. The external jugular vein is easier to visualize and studies have demonstrated that this is a reliable method that correlates highly with catheter measured CVP.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years or older at the time of enrolment
* Chronic Kidney Disease patients and healthy volunteers
* Participants should be able to provide written informed consent
* Subject is termed eligible as determined by Pre-Screening Phase (as defined in protocol)

Exclusion Criteria:

* Unable to identify external jugular vein (EJV)
* Unable to identify internal jugular vein (IJV)
* Unable to access right side of subject's neck
* Allergic to adhesive tape
* History of central vein stenosis
* Undergoing photodynamic therapy (PDT)
* Presence of an arteriovenous fistula

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Adult patients with Chronic Kidney Disease (CKD)
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)

PRIMARY OUTCOMES:
Central Venous Pressure (CVP) | 0-3 hours
  To determine if the CVP from the non-invasive monitor correlates with the CVP from physical examination

CONTACTS AND LOCATIONS:
Overall Officials: Azim S Gangji, MD, Principal Investigator — St. Joseph's Healthcare Hamilton; Melissa T Perri, MESc, Study Director — Mespere Lifesciences Inc.
Locations (1):
- St. Joseph's Hamilton Healthcare, Hamilton, Ontario, Canada